CLINICAL TRIAL: NCT04006717
Title: Evaluation of Post-Endodontic Pain Control Using Low- Level Laser Therapy in Comparison to Intra-canal Cryotherapy: a Randomized Placebo-controlled Clinical Trial
Brief Title: Comparison Between Low-level Laser Therapy, Intracanal Cryotherapy and Their Combination, on Post-endodontic Pain Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Ibrahim Khalaf, Assistant Professor, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MisrIU
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2023-02

CONDITIONS: Low-level Light Therapy; Cryotherapy
Keywords: Post-endodontic pain; Low-level laser; Intracanal cryotherapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (No Intervention): Routine root canal treatment
- Low-Level Laser Placebo (Placebo Comparator): Patient informed that laser will be applied but device won't be turned on
  Interventions: Device: Low Level Laser therapy
- Low-Level Laser Therapy (Experimental): Low-Level Laser Therapy following root canal treatment
  Interventions: Device: Low Level Laser therapy
- Intracanal Cryotherapy (Experimental): Cold saline irrigation before obturation
  Interventions: Procedure: Intra canal Cryotherapy
- Combination of LLLT and ICCT (Experimental): Both cold saline irrigation before obturation and Low-level laser Therapy after root canal treatment
  Interventions: Device: Low Level Laser therapy; Procedure: Intra canal Cryotherapy

INTERVENTIONS:
Device: Low Level Laser therapy — Diode laser (EPIC™ BIOLASE) with wavelength 940nm
  Arms: Combination of LLLT and ICCT; Low-Level Laser Placebo; Low-Level Laser Therapy
Procedure: Intra canal Cryotherapy — Irrigation with cold saline 2-4 C
  Arms: Combination of LLLT and ICCT; Intracanal Cryotherapy

SUMMARY:
Statement of the problem: Postoperative pain following endodontic treatment is a common complication that might require analgesics for pain relief. Low-level laser therapy (LLLT) and Intracanal Cryotherapy (ICCT) are both recommended as non-pharmacological and non-invasive treatment modalities for management of painful situations. Aim of the study: This study is conducted to clinically evaluate and compare the effect of both LLLT and ICCT on post-endodontic pain (PEP) over 5 days in molars with symptomatic apical periodontitis (SAP) using visual analog scale (VAS). Materials & Methods: This parallel arm, randomized clinical trial will involve 95 systemically free patients with SAP in molars. The patients will be randomly allocated to 5 equal groups as follows: control (no intervention), placebo (mock laser therapy), LLLT, ICCT and a combination of both. Postoperative pain levels after 6 hrs, 12 hrs, on 2nd day and 5th day are going to be assessed on the VAS and shall be noted. Data collected will be tabulated and statistically analysed.

DETAILED DESCRIPTION:
Selection of patients:

Ninty-five patients shall be selected from the regular pool of patients visiting Misr International University Dental Clinic Complex. After application of inclusion and exclusion criteria, preoperative and percussion pain shall be recorded on a 10-cm VAS by the patients. Percussion will be performed by tapping on the occlusal surfaces of the teeth with the back of a mirror handle. It will be assessed prior to the root canal treatment by the operator who shall be performing the root canal treatment. Diagnosis of the tooth as symptomatic apical periodontitis will be done according to the book Cohen's Pathways of the Pulp. Clinical symptoms are going to be defined as follows:

1. Severe preoperative pain (VAS >6)
2. Severe percussion pain (VAS > 6) Patients with all inclusion criteria will be offered to participate in the study.

Grouping of samples:

Each selected patient will get a unique serial code that is previously distributed among the 5 groups randomly. Nineteen patients in each as follows; Group 1: Control (no intervention), Group 2: Placebo (mock laser therapy), Group 3: LLLT, Group 4: ICCT and Group 5: Combination of both LLLT and ICCT. New patients will be incorporated in the study in place of lost patients.

Method:

After the patient signs the attached consent form, profound anesthesia and rubber dam application shall be ensured. Standard chemo-mechanical preparation parameters (Master Apical File: size #25 to #40 k-files depending on anatomical features of the roots) shall be followed. Obturation will be performed using lateral compaction technique. In Group 4 and Group 5, cold saline with temperature ranging from 2-4 °C, will be used as a final rinse using a conventional syringe. LLLT using diode laser (EPIC™ BIOLASE) with wavelength 940nm will be applied towards the tissues surrounding the roots of treated molars in Group 3 and 5 after completing obturation and sealing the access cavity. In Group 2, the diode laser tip shall be placed at approximately 10 mm from the tissue around the apices of the treated roots; however, it won't be activated.

Data collection:

All patients will be instructed to complete a survey at home. Pain is going to be evaluated based upon a questionnaire filled by the patient after 6 hrs, 12 hrs, on 2nd day and 5th day after root canal treatment. Any of the patients taking analgesics after the treatment, shall be advised to note this in the questionnaire. The information collected from the questionnaires covers the occurrence and the intensity of PEP. The intensity of pain will be evaluated on a numeric rating scale (VAS) of 0 for "no pain" to 10 for "unbearable pain". Patients will return the filled questionnaire on the 5th day after treatment and they shall be assured via telephone contact.

Blinding:

Outcome assessors and statistician will be blinded. Both the participants and principal investigators can't be blinded owing to the use of two obviously different methods, LLLT and ICCT or no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a molar tooth with symptomatic apical periodontitis indicated for root canal treatment.
* Systemically free patients. ASA I
* Teeth with mature apex.
* Teeth without root resorption.

Exclusion Criteria:

* Patients with other pulpal diagnoses.
* Medically compromised patients.
* Pregnant females.
* Patients taking analgesics or anti-inflammatory drugs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Post-endodontic pain | 5 days
  Score on Visual Analogue scale, ranging from 1 (No pain) to 10 (Worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No